CLINICAL TRIAL: NCT01207245
Title: Circadian Rhythm In Tobramycin Elimination In Cystic Fibrosis (CRITIC) A Randomized Pharmacokinetic Comparison of Tobramycin in Cystic Fibrosis
Brief Title: Circadian Rhythm In Tobramycin Elimination In Cystic Fibrosis
Acronym: CRITIC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10076; NIHR RfPB PB-PG-1207-15025 (Other Grant/Funding Number: National Institute of Health Research)
Record Dates: First submitted 2010-09-21; First posted 2010-09-22 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; Tobramycin; Pharmacokinetics; Toxicity
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Morning dose of tobramycin (Active Comparator): Administration of tobramycin once daily dose in the morning
  Interventions: Other: Tobramycin time of administration
- Evening tobramycin (Active Comparator): Evening dose of tobramycin once daily
  Interventions: Other: Tobramycin time of administration

INTERVENTIONS:
Other: Tobramycin time of administration — Random allocation to time of day of administration of tobramycin

SUMMARY:
Cystic fibrosis is the most common inherited life limiting condition which affects children. Patients with it develop lung infections which become difficult to clear, and damage the lungs. These are treated with antibiotics (such as tobramycin) into the vein (termed "intravenous antibiotics"). This has without doubt improved survival. However, all treatments have side effects. Tobramycin can cause kidney damage. The investigators have preliminary data that suggests that administering tobramycin in the morning may be safer for the kidneys than administering it in the evening.

The investigators plan to approach children and adults with cystic fibrosis whose doctors have decided to administer a course of intravenous tobramycin. The investigators will randomly allocate them to receive it at either 0800h or 2200h. The investigators will measure the rate at which the body eliminates tobramycin from the bloodstream, by measuring the amount of tobramycin in the blood stream after administering the antibiotic. For each patient the study will last for the duration of the course of antibiotics. This is decided by the doctor looking after the patient (rather than the researcher), and would typically be 14 days. The investigators will also measure substances in the blood and urine ("biomarkers") which are sensitive indicators of low levels of kidney injury. The investigators will monitor lung function and lung bacteria in both the groups to ensure that the patients in both groups improve by the same amount.

If the preliminary data are proved correct, this research will allow investigators to improve the safety profile of tobramycin, one of the most widely prescribed drugs in cystic fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cystic fibrosis (CF) (defined as clinical features of CF plus a positive sweat test OR the presence of 2 genes known to be associated with CF disease)
* Males or female 5 years and older
* Treating doctor has decided to commence a course of tobramycin
* Patient or parent / legal guardian able to give informed consent

Exclusion Criteria:

* Previous episode of acute kidney injury
* Solid organ transplantation
* Evidence of impaired renal function (raised serum creatinine above the normal range for age)
* Once daily aminoglycoside unsuitable because of hypersensitivity or previous high trough levels on once daily dosing.
* Pregnancy

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-05; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Renal Elimination Rate Constant of Tobramycin | Days 1, 8 and 14

SECONDARY OUTCOMES:
Weight | Day 1, 8, 14
Pulmonary Function | Day 1, 8, 14
Urinary Biomarkers | Days 1 and 14
  NAG, NGAL, IL-18, KIM1, Cystatin C
Serum biomarkers | Days 1 & 14
  Serum creatinine Serum Cystatin C Estimated GFR
Serum Electrolytes | Days 1 & 14
  Serum Potassium and Magnesium

CONTACTS AND LOCATIONS:
Overall Officials: Alan Smyth, Principal Investigator — University of Nottingham
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, Nottinghamshire, United Kingdom

REFERENCES:
- [Derived] Prayle AP, Jain K, Touw DJ, Koch BC, Knox AJ, Watson A, Smyth AR. The pharmacokinetics and toxicity of morning vs. evening tobramycin dosing for pulmonary exacerbations of cystic fibrosis: A randomised comparison. J Cyst Fibros. 2016 Jul;15(4):510-7. doi: 10.1016/j.jcf.2015.07.012. Epub 2015 Aug 15. PMID 26282839